CLINICAL TRIAL: NCT03500523
Title: Corneal Biomechanical Properties in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Funda Dikkaya, principal investigator, Medipol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 11134
Record Dates: First submitted 2018-04-03; First posted 2018-04-18 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Corneal Biomechanics; Pregnancy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1-study group (Experimental): study group: pregnant women
  Interventions: Diagnostic Test: corneal biomechanical properties
- 2-control group (Experimental): control group: healthy non pregnant women
  Interventions: Diagnostic Test: corneal biomechanical properties

INTERVENTIONS:
Diagnostic Test: corneal biomechanical properties — We want to investigate changes of corneal biomechanical properties during pregnancy. The Ocular Response Analyzer (ORA) evaluate the in vivo corneal biomechanical properties in form of corneal hysteresis (CH) and corneal resistance factor (CRF)

SUMMARY:
57 eyes of 57 healthy pregnant women who were visiting Obstetrics and Gynecology department for routine examination and 26 eyes of 26 non pregnant control subjects who were at the first week of the menstrual cycle were enrolled in the study. All subjects had a detailed ophthalmologic examination including the best corrected visual acuity with a Snellen chart, slit- lamp biomicroscopic evaluation, and indirect fundoscopy. The biomechanical properties Corneal Hysteresis, Corneal resistance factor, corneal compensated intraocular pressure and Goldmann-correlated intraocular pressure values were measured with ORA (Ocular Response Analyzer, software version 1.02, Reichert, Inc.) Central corneal thickness was measured with a built-in ultrasonic pachymeter attached to the ORA device.Axial length , Anterior chamber depth , and keratometry readings were acquired with an ocular biometer (IOLMaster; Carl-Zeiss Meditec, Inc.) before CCT determinations had been taken. Results of these parameters were compared between pregnant group and healthy control group.

ELIGIBILITY:
Inclusion Criteria:

* 57 eyes of 57 healthy pregnant women who were visiting Obstetrics and Gynecology department for routine examination and 26 eyes of 26 non pregnant control subjects who were at the first week of the menstrual cycle were included in the study.

Exclusion Criteria:

* Exclusion criteria included history of intraocular surgery or refractive surgery, history of glaucoma or glaucoma suspicion, contact lens wear, systemic autoimmune disease or diabetes and usage of eye drop and oral contraceptives.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 83 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-03-31 (Actual); Study Completion 2018-03-31 (Actual)

PRIMARY OUTCOMES:
changes of corneal hysteresis during pregnancy | three months
  we analyzed the biomechanical properties of the cornea in terms of corneal hysteresis (mmHg) by using ocular response analyzer device in healthy pregnant women and compared the data with non pregnant women.
changes of corneal resistance factor during pregnancy | three months
  we analyzed the biomechanical properties of the cornea in terms of corneal resistance factor (mmHg) by using ocular response analyzer device in healthy pregnant women and compared the data with non pregnant women.

CONTACTS AND LOCATIONS:
Locations (1):
- Funda Dikkaya, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No